CLINICAL TRIAL: NCT05006014
Title: Primary Versus Secondary Implant Stability in Relation to Gap Distance of Immediate Implant With Immediate Loading by Provisional Restoration
Brief Title: Immediate Implant With Provisionalization
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Dalya Munther Naeem, Bachelor of dental surgery ( master student ), University of Baghdad
Other Study IDs: 1427705
Record Dates: First submitted 2021-08-04; First posted 2021-08-16 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Maintain the Esthetic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Patient with non restorable teeth: Patient with non restorable teeth located in smile line needs extraction with immediate implantation and immediate provisionalization to improve psychiatric effect of tooth loss
  Interventions: Procedure: Tooth guided immediate implant placement

INTERVENTIONS:
Procedure: Tooth guided immediate implant placement — The technique of implant insertion consisted of a progressive preparation of the implant site using the anatomy of the root of the single rooted teeth to be extracted as a reference and as aid for apical engagement

SUMMARY:
Prospective observational clinical study conducted to evaluate the success of graftless immediate implantation with provisionalizaion

DETAILED DESCRIPTION:
In this study 35 graftless immediately placed implant in smile line loaded by provisional office made restoration, the primary and secondary stability measured and compared in addition to evaluation of pink esthetic score

ELIGIBILITY:
Inclusion Criteria:

1. Medical and psychological fitness for minor oral surgery.
2. Age 20-60 years.
3. medium to thick gingival biotype.
4. buccal plate thickness more than (1mm).

Exclusion Criteria:

1. Smoking habit.
2. Diabetes mellitus.
3. A systemic disorder that is contraindicated for the minor surgical procedure.
4. Pregnancy or lactation.
5. Any irradiation in head and neck area.
6. Need for bone augmentation procedure.
7. Clinical signs of bruxism or other severe functional disorders.
8. patient with periodontal disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adult with non restorable dental unit seeking for immediate implantation with provisionalization
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2021-01-27 (Actual); Primary Completion 2021-11-27 (Actual); Study Completion 2022-03-27 (Estimated)

PRIMARY OUTCOMES:
Implant primary stability | 0 day
  The stability measured by resonance frequancy analysis device (osstell)
Jumping gab | 0 day
  The gab that located between the implant surface and buccal plate
Pink esthetic score | 0 day, before extraction and implant placement
  Denote the esthetic profile of bone and gingiva

SECONDARY OUTCOMES:
Implant secondary stability | Up to 16 weeks
  The stability measured by resonance frequancy analysis device (osstell)
Ridge reduction | Up to 16 weeks
  The amount of reduction in buccal profile of the alveolar ridge
Pink esthetic score | after implantation By 4 months
  Denote the esthetic profile of bone and gingiva

CONTACTS AND LOCATIONS:
Locations (1):
- College of dentistry, Baghdad, Bab Al Moatham, Iraq